CLINICAL TRIAL: NCT03424135
Title: An Open Label Crossover Pharmacokinetic Trial of Naproxen Sodium and Diphenhydramine Hydrochloride Soft Capsules Versus Naproxen Sodium and Diphenhydramine Hydrochloride Tablets in Healthy Adult Subjects Under Fed Conditions
Brief Title: A Pharmacokinetic Trial of Naproxen Sodium and Diphenhydramine Hydrochloride Soft Capsules Versus Naproxen Sodium and Diphenhydramine Hydrochloride Tablets in Healthy Adult Subjects Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17944
Record Dates: First submitted 2018-02-01; First posted 2018-02-06 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Clinical Pharmacology
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test product + Reference product (Experimental): Each treatment sequence consists of two treatment periods (Dosing Periods 1 and 2) with each period consisting of 4 days starting with an overnight fast of at least 10 hours. Subjects will consume a standardized high calorie, high fat breakfast approximately 30 minutes prior to dosing followed by a single dose of study drug administration the morning of Day 1, then a 72-hour PK blood sampling period. The two study drug administrations are separated by a 7 calendar days washout phase.
  Interventions: Drug: Naproxen sodium and diphenhydramine hydrochloride soft capsules; Drug: Naproxen sodium and diphenhydramine hydrochloride coated tablets (Aleve PM, BAY98-7111)
- Reference product + Test product (Experimental): Each treatment sequence consists of two treatment periods (Dosing Periods 1 and 2) with each period consisting of 4 days starting with an overnight fast of at least 10 hours. Subjects will consume a standardized high calorie, high fat breakfast approximately 30 minutes prior to dosing followed by a single dose of study drug administration the morning of Day 1, then a 72-hour PK blood sampling period. The two study drug administrations are separated by a 7 calendar days washout phase.
  Interventions: Drug: Naproxen sodium and diphenhydramine hydrochloride soft capsules; Drug: Naproxen sodium and diphenhydramine hydrochloride coated tablets (Aleve PM, BAY98-7111)

INTERVENTIONS:
Drug: Naproxen sodium and diphenhydramine hydrochloride soft capsules — Single oral administration of Naproxen sodium 220 mg/DPH HCl 25mg (2 capsules)
Drug: Naproxen sodium and diphenhydramine hydrochloride coated tablets (Aleve PM, BAY98-7111) — Single administration of Naproxen sodium 220 mg/DPH HCl 25mg (2 tablets)

SUMMARY:
To evaluate the relative bioavailability of naproxen sodium/diphenhydramine hydrochloride (DHP HCL) 220/25 mg soft capsules (Test) versus naproxen sodium/DPH HCl 220/25 mg tablets (Reference) after a single oral administration (2 x naproxen sodium 220 mg and DPH HCl 25 mg combination product) under fed conditions in healthy adult subjects.

To assess the safety and tolerability of the investigational products in terms of adverse events (AEs) and clinical parameters (systolic/diastolic blood pressure, pulse rate, physical examination, clinical and laboratory testing).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory male and female subjects between 18 to 55 years of age inclusive;
* Body Mass Index (BMI) in the range of 18 to 30 kg/m2 inclusive; and a total body weight >50 kg (110 lbs.);
* Results of screening and clinical laboratory tests are within normal range or considered not clinically significant by the Principal Investigator and Sponsor;
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives) [e.g., hormonal contraceptives (oral, patch, injectable or vaginal ring), implantable device (implantable rod or intrauterine device), or a double barrier] and have a negative pregnancy test at Screening and prior to study drug administration on Day -1 of Dosing Periods 1 and 2. Female subjects of non-childbearing potential must be amenorrheic for at least two years or have had a hysterectomy and/or bilateral oophorectomy;

Exclusion Criteria:

History of hypersensitivity symptoms with the use of naproxen/naproxen sodium, diphenhydramine hydrochloride/citrate, acetylsalicylic acid (ASA), other Nonsteroidal anti-inflammatory drugs (NSAIDs) or similar pharmacological agents or components of the products;

* Females who are pregnant or lactating;
* Vegetarian or restricted diet (e.g., gluten-free);
* Any active disease, acute or chronic;
* Have taken naproxen/naproxen sodium, DPH HCl or diphenhydramine citrate, DPH HCl or diphenhydramine citrate-containing products, acetylsalicylic acid, ASA-containing products, acetaminophen, ibuprofen, any other NSAIDs (Over-the-Counter [OTC] or prescription) or NSAID containing products, xanthines, antihistamines or caffeine-containing products (e.g., coffee, tea and chocolate) 7 days prior to dosing or during the Dosing Periods, other than trial treatment;
* Use of any over-the-counter or prescription medications, vitamins or herbal supplements (except acceptable forms of birth control) within 7 days prior to dosing or throughout the trial, unless in the opinion of the Investigator, the medication will not interfere with the trial procedures, data integrity, or compromise the safety of the subject;
* Positive test for Human immunodeficiency virus (HIV) antibodies and antigens;
* Positive test for hepatitis B surface antigen (HBsAg) test;
* Positive test for anti-hepatitis C virus (Anti-HCV) antibodies;
* In the judgment of the investigator, any need of other medication during the trial besides the test and reference study medication;
* Recently had (past 30 days) or plan to have surgery, an invasive procedure, tattoos or piercings during the trial or within 2 weeks after treatment;
* More than moderate alcohol consumption (>40 g of alcohol regularly per day);
* Positive alcohol or drug screen at Screening or on Day -1 of each dosing period.
* Any history or suspicion of barbiturate, amphetamine, benzodiazepine, cocaine, opiates, methamphetamine or cannabis abuse;
* Loss of blood in excess of 50 mL to 499 mL within 30 days or 500 ml or greater within 56 days of the first dose of trial treatment (e.g., donation, plasmapheresis or injury);
* Excessive sports or sauna within 5 days before start of the treatment phase and willing to abstain during the trial;
* Have a platelet count <150,000/mm3 and in the judgment of the investigator, presents a significant bleeding risk;
* History of gastrointestinal bleeding or perforation, related to previous NSAID therapy. Active, or history of recurrent peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding);
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary (including emphysema and chronic bronchitis), gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases, (including glaucoma or benign prostatic hypertrophy) or malignancies or any disease or condition which could influence the metabolism of the drug;
* Smokers or currently consuming any type of tobacco product(s) including any smoking cessation nicotine-containing product within the previous three months (e.g., nicotine patch, nicotine gum);
* Not willing to abstain from any xanthine-containing or grapefruit/ pomelos -containing food/beverages during the study;
* Have a previous medical history of gout or reduced uric acid excretion;
* Alcoholism or drug abuse within 2 years prior to the Screening Visit;
* Consumed alcohol within 24 hours prior to dosing of investigational medicinal product (IMP) in the study center on study days (verified by saliva/breath alcohol test on Day -1 of each Dosing Period);
* Current or past history of controlled substance dependence;
* Current participation in any other trials involving investigational or marketed products within 30 days prior to the Screening Visit;
* Member or relative of study staff or the Sponsor directly involved in the study;
* Unwilling or unable to comply with all requirements outlined in the protocol
* Subjects with a medical disorder, condition, or history of such that could impair the subject's ability to participate or complete this trial in the opinion of the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
AUC | Within 30 minutes prior to dosing (baseline) 20, 40, 60 minutes and 1 h 30 min, 2 h, 2 h 20 min, 2 h 40 min, 3, 3 h 20 min, 3 h 40 min, 4 h, 4 h 30 min, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose.
  Area under the concentration vs. time curve from zero to infinity after single (first) dose
AUC(0-tlast) | Within 30 minutes prior to dosing (baseline) 20, 40, 60 minutes and 1 h 30 min, 2 h, 2 h 20 min, 2 h 40 min, 3, 3 h 20 min, 3 h 40 min, 4 h, 4 h 30 min, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose.
  Area under plasma concentration vs. time curve from zero to last data point >LLOQ (lower limit of quantitation), calculated up by linear trapezoidal rule, down by logarithmic trapezoidal rule
Cmax | Within 30 minutes prior to dosing (baseline) 20, 40, 60 minutes and 1 h 30 min, 2 h, 2 h 20 min, 2 h 40 min, 3, 3 h 20 min, 3 h 40 min, 4 h, 4 h 30 min, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose.
  Maximum observed drug concentration, directly observed from analytical data

SECONDARY OUTCOMES:
Number of adverse events as a measure of safety and tolerability | Up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- ICON Development Solutions, LLC, San Antonio, Texas, United States